CLINICAL TRIAL: NCT01956461
Title: Effects of Teriparatide Therapy for Japanese
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tomidahama Hospital (Other)
Responsible Party: Principal Investigator, Toshihiko Kono, Head of Hospital, Tomidahama Hospital
Other Study IDs: IRB TH No 6
Record Dates: First submitted 2013-09-21; First posted 2013-10-08 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Osteoporosis
Keywords: osteoporosis; BMD; teriparatide; nursing home
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
In this study, the investigators would like to analyze the bone mineral density (BMD) , bone turnover makers, and fracture prevention effects of daily teriparatide in Japanese patients under clinical practice. The participants are treated in the investigators hospital, who are under severe osteoporotic condition.

Several determinants were reported to be related to subsequent BMD increase, such as baseline bone turnover markers (BTMs), low BMD at baseline, age, prior treatment, but comprehensive discussion is lacking. Specifically, there analyses were performed fragmentarily.

The main objective of this study is to reveal the determinants of subsequent BMD increase and fracture preventing effect by teriparatide.

Next, in Japan, as the baby boom generation retires, aging and depopulation occur rapidly. As a result, there is a lot of nursing home. But there are few reports concerning to the efficacy of teriparatide treatment in nursing home patients. The second objective is to reveal the efficacy of teriparatide for patients living nursing home, especially BMD changes, bone turnover makers change, and adverse events.

DETAILED DESCRIPTION:
Registry criteria: Patients treated in the investigators hospital using teriparatide. Enrolled patients are severe osteoporosis; more than two previous osteoporotic fractures, low BMD (< young adult mean 65%).

Interventions: blood analyses and dual-energy X-ray absorptiometry (DXA) every 4 months Informed consent: Written informed consent will be obtained. Sample size: Five-hundreds participants

ELIGIBILITY:
Inclusion Criteria:

* severe osteoporotic patients

Exclusion Criteria:

* cancer, hypercalcemia, etc (i.e. patients who could not use teriparatide)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Osteoporotic patients who admit to our hospital
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2010-09; Primary Completion 2016-11 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
The determinants related to BMD increase and fracture prevention for teriparatide treatment | Up to 36 months
  The investigators plan to analyze 500 patients who undergo teriparatide treatments 12 months. To enroll 500 participants, up to 24 months is required beside 12 months treatment periods.
  We investigate several determinants related to BMD increase, such as baseline age, gender, body mass index, BMD, BTMs, history of fracture, and prior treatment. We also investigate determinants related to fracture prevention effects by teriparatide treatment, such as baseline age, gender, body mass index, BMD, BTMs, history of fracture, prior treatment, walking ability, dementia,and site of living.
  To determine the response variables of BMD changes and fracture prevention effects, initially univariate analyses are performed by Spearman correlation coefficients and Mann-Whitney U test. Data are further analyzed with a multiple regression. To estimate odds ratios and 95% confidence intervals (95% CIs) of each determinants, logistic regression analyses are performed.

SECONDARY OUTCOMES:
BMD and BTMs response, and fracture prevention effects of teriparatide for the patients in nursing home | Oct 2014
  We plan to evaluate longitudinal BMD and BTMs changes for 24 months. BMD was evaluated every four months, ans BTMs are evaluated one months after treatment, and every four months. Fracture prevention effects are evaluated by radiography, if fracture is suspected. Statical analyses are performed using Spearman correlation coefficients, paired t-test, Mann-Whitney U test, and Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Locations (1):
- Tomidahama Hospital, Yokkaichi, Mie-ken, Japan